CLINICAL TRIAL: NCT04955392
Title: Effects of an Osteopathic Treatment Protocol on Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramón Mateos Alpuente (Other)
Responsible Party: Sponsor-Investigator, Ramón Mateos Alpuente, Principal Investigator, Ramon Mateos Fisioterapia y Osteopatía
Organization: Ramon Mateos Fisioterapia y Osteopatía (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SQ001
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Sleep Disorder
Keywords: Sleep quality; Heart Rate Variability; Stress; Osteopathic Manipulative Treatment; Manual Therapy
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: SIngle-centre interventional single-blinded randomized contsubjectsrolled trial, with random assignment of the subjects in two groups (intervention and control, 1: 1 ratio)
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible and recruited patients will be Randomized using OxMaR software (Oxford Minimization and Randomization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group of patients that will receive the 4 techniques proposed to evaluate the changes on sleep quality
  Interventions: Other: Osteopathic treatment protocol
- Control group (Sham Comparator): Group of patients that will receive a sham technique
  Interventions: Other: Sham technique

INTERVENTIONS:
Other: Osteopathic treatment protocol — The intervention protocol consists of 4 techniques that will be performed according to the following order:
  1. Inhibition of the suboccipital muscles.
  2. Parietal Lift.
  3. Sutherland Technique of Sphenobasilar Synchondrosis.
  4. Compression technique of the fourth ventricle (CV4).
  Arms: Intervention group
Other: Sham technique — Sham technique that consists of placing the hands on top of the skull without any therapeutic intention for five minutes.
  Arms: Control group

SUMMARY:
SIngle-centre interventional single-blinded randomized controlled trial, with random assignment of the subjects in two groups (intervention and control, 1: 1 ratio) and to be carried out with volunteers that present alterations in the quality of sleep. Eligible and accepting subjects participating in the study will be assigned to receive an osteopathic treatment protocol or a placebo technique

DETAILED DESCRIPTION:
Intervention protocol in the intervention group:

The intervention protocol consists of 4 techniques that will be performed according to the following order:

1. Inhibition of the suboccipital muscles.
2. Parietal Lift.
3. Sutherland Technique of Sphenobasilar Synchondrosis.
4. Compression technique of the fourth ventricle (CV4).

Intervention protocol in the control group:

Placebo technique that consists of placing the hands on top of the skull without any therapeutic intention for five minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults ranging from 18 to 80 years old and with a score greater than 5 on the Pittsburgh Sleep Quality Index

Exclusion Criteria:

1. Recent head injuries or fractures.
2. Having suffered a stroke or intracranial hemorrhage.
3. Tumors.
4. Epilepsy.
5. Bradycardia.
6. Hypotension.
7. Heart disease
8. Neurological problems
9. Psychiatric problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 1 month
  Sleep quality is measured using the Pittsburgh Sleep Quality Index before the intervention and one month after, having received three treatment sessions.

SECONDARY OUTCOMES:
Heart Rate Variability | 1 month
  Changes in Heart Rate Variability (HRV) that will be measured and monitored before and at the end of the intervention using a portable HRV monitoring device (polar H10) that sends the signal to a computer for its collection and analysis through the Kubios HRV software
Perceived Stress | 1 month
  Assessment of perceived stress using the Cohen's Perceived Stress Scale (PSS), which will be completed before the first intervention and one week after completing the three planned interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Mateos Alpuente, Principal Investigator
Locations (1):
- Ramón Mateos Fisioterapia y Osteopatía, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No